CLINICAL TRIAL: NCT02180347
Title: Contact Lenses and Myopia
Acronym: CLAM
Status: Completed | Type: Observational
Sponsor: State University of New York College of Optometry (Other)
Responsible Party: Principal Investigator, Kathryn Richdale, Assistant Professor, State University of New York College of Optometry
Other Study IDs: CLAM_602929; CLAM_602929 (Other: SUNY College of Optometry)
Record Dates: First submitted 2014-06-30; First posted 2014-07-02 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Myopia
Keywords: Pediatrics; Contact lenses
MeSH Terms: conditions — Myopia | interventions — Contact Lenses

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Multifocal contact lenses: Coopervision Proclear Multifocal
  Interventions: Device: Contact lenses
- Single vision contact lenses: Coopervision Proclear Sphere
  Interventions: Device: Contact lenses

INTERVENTIONS:
Device: Contact lenses

SUMMARY:
The objective of this study is to determine if multifocal contact lenses affect accommodation and/or binocular vision when worn by pediatric patients. This will be accomplished through subjective and objective accommodative and binocular experiments in children wearing single vision and multifocal soft contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* 7 to 15 years of age
* Refractive error between -1.00 and -8.00 D sphere, with less than or equal to 1.00 D astigmatism
* Corrected visual acuity of 20/25 or better in each eye

Exclusion Criteria:

* Ocular or systemic disease known to affect accommodation or vision
* Convergence or accommodative disorder, or any strabismus
* Use of oral or topical medications known to affect accommodation

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population includes children and teens that are recruited from the University Eye Center at SUNY College of Optometry and from the greater New York City area.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2014-06; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Accommodative response | Up to two hours
  Accommodative response will be measured subjectively and objectively using the push-up technique and photorefraction.
Binocular posture status | Up to two hours
  Binocular posture will be measured using Modified Thorington,

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Richdale, OD, PhD, Principal Investigator — State University of New York College of Optometry
Locations (1):
- SUNY College of Optometry, Clinical Vision Research Center, New York, New York, United States